CLINICAL TRIAL: NCT06417541
Title: Autopsy and Photon Counting Computed Tomography to Evaluate Thromboses Related to Central Venous Catheters (PHOTO CAT)
Brief Title: Autopsy and Photon Counting Computed Tomography to Evaluate Thromboses Related to Central Venous Catheters
Acronym: PHOTO CAT
Status: Recruiting | Type: Observational
Sponsor: Thomas Kander (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Sponsor investigator, Region Skane
Organization: Region Skane (Other)
Other Study IDs: PHOTO CAT
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Central Venous Catheter Thrombosis
Keywords: central venous catheter; thrombosis; photon counting ct
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Thrombosis | interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased patients with an indwelling central venous catheter: Sub study 1, Diseased patients with an indwelling central venous catheter
  Interventions: Diagnostic Test: Diseased patients with an indwelling central venous catheter who is referred to autopsy
- Living patients with an indwelling central venous catheter: Living patients with an indwelling central venous catheter who are referred to a CT-scan without intravenous contrast
  Interventions: Radiation: Living patients with an indwelling central venous catheter referred to a CT scan without iv contrast

INTERVENTIONS:
Diagnostic Test: Diseased patients with an indwelling central venous catheter who is referred to autopsy — Photon counting CT is performed and the results are compared to the results of the autopsy
  Groups: Diseased patients with an indwelling central venous catheter
Radiation: Living patients with an indwelling central venous catheter referred to a CT scan without iv contrast — Patients will be investigated using a photon counting CT. Prior to the investigation patients will be investigated with ultrasound. The results from the two modalities will be compared
  Groups: Living patients with an indwelling central venous catheter

SUMMARY:
Central venous (CVC) is essential in modern healthcare but unfortunately associated with complications, including thrombosis. In a recently published study, it was showed that 12 out of 12 deceased patients had subclinical CVK-related thrombosis (Rockholt et al.). To shed light on this problem, the current studies were designed. In sub-study 1, deceased patients with CVC who are referred for clinical autopsy are included. Before the autopsy, the deceased will be examined with a photon-counting computed tomography (CT) scan and the results will be compared.

In sub-study 2, living patients with CVC who are referred for various CT scans without contrast, are included. After informed consent, the patient will be examined with the photon-counting CT, whose reliability has been validated in Part 1 and the incidence of subclinical CVC-related thrombosis will be reported.

DETAILED DESCRIPTION:
Purpose and specific objective The aim of the current project (PHOTO CAT) is to evaluate the prevalence of subclinical thromboses related to central venous catheters (CVCs) using a novel high-resolution photon-counting computed tomography (CT) scan and to evaluate the performance of the photon-counting CT compared to clinical autopsy.

Scientific questions

1. Can the photon-counting CT diagnose subclinical CVK-related thromboses detected at later autopsy?
2. How common are CVC-related thromboses in autopsies of deceased people with existing CVC?
3. How does the performance of the photon counting DT compare to clinical autopsy?
4. How common are CVC-related thromboses in a cohort that does photon-counting DT for various reasons and has a CVC?
5. Can imaging be improved by adjustments to the DT protocol?
6. Can an ultrasound scan on living patients diagnose subclinical CVK-related thrombosis detected by photon-counting CT?

Background CVCs are essential in modern healthcare and have a wide range of applications. They enable direct access to the central bloodstream and are used, among other things, to administer medicines, nutrition and to monitor blood circulation. Unfortunately, they are associated with a variety of complications, including thrombosis. Studies report thrombosis incidences between 5 - 30% in living patients. When the CVC is introduced into the blood vessel, a number of physiological defense systems are initiated. Inflammation and clotting are activated, leading to the formation of a fibrin stocking around the catheter. This can then develop into a catheter-related thrombosis, which in turn can have serious consequences for the patient, such as pulmonary embolism or infection.

Photon-counting DT is the new generation of DT. What distinguishes this from the traditional one is that the radiation through the body is detected with a new type of detector that measures each X-ray, which provides significantly greater precision and resolution for a given radiation dose compared to traditional CT. This is particularly valuable in imaging diagnostics that rely on detailed morphology such as high-resolution CT of lungs. In order to achieve its full potential with as little radiation dose and contrast volume as possible with preserved image resolution, the design of protocols for the photon-counting CT needs to be optimized.

Autopsy studies on CVC-related thrombosis and vascular changes are few. In a case series from 1994, changes in the vessel wall were examined macroscopically and biofilms were assessed with electron microscopy. The presence of fibrin stocking on the surface of all CVCs (n = 72), and wall-mounted thrombosis was reported in 38% of cases. In another autopsy study, Forauer et al. demonstrated severe CVC-related vascular changes that included intima damage with infiltration of media by inflammatory cells and varying degrees of adherent thrombus. Wichmann et al. published data showing a 38% prevalence of macroscopic catheter-related thrombosis in 61 human autopsies. In a recently published autopsy study, we showed that 12 out of 12 cases had CVC-related mural thrombosis at autopsy, with most being located in the distal part of the CVC (Rockholt et al.).

There are also a number of clinical studies that have investigated how common CVC-related thrombosis is using ultrasound. In a well-designed prospective study, 16.9% of ICU patients had subclinical CVK-related thrombosis. The problem with the ultrasound method is that the distal part of the CVC is difficult to visualize with ultrasound, which means that the thrombosis incidence risks being underestimated.

Material and method In an attempt to investigate how common subclinical CVK-related thrombosis, the current studies, include photon-counting CT, were designed.

In substudy 1, photon counting CT is used to examine deceased intensive care patients referred for autopsy on clinical indication, with CVC in-situ. The CT will be focused on the vein with the CVC but a full body examination will also be done . Both examination results will be compared with the clinical autopsy conducted after the examinations. This first part of PHOTO CAT includes Scientific questions 1-3.

In sub-study 2, living patients with CVC who are referred for CT scan without contrast, will be eligable for inclusion. After consent, the study will be carried out with photon counting CT in two phases. First, the examination for which the patient was referred, will be performed. In the second phase, a targeted examination is performed for research purposes of the vein with the CVC. Within 12 hours before or after the CT scan, it is planned to perform an ultrasound scan of the vein where the CVC is located. The aim is to evaluate the performance of ultrasound examination in detecting CVC-related thrombosis, compared to photon-counting CT. Sub-study 2 of PHOTO CAT includes Questions 4-6.

Analysis of data and statistics No one has previously reported photon-counting CT to detect CVC-related thromboses. Therefore, the current exploratory study is planned. The results may form the basis for sample size calculation in future studies.

Significance In patients with CVC, subclinical CVC-related thromboses are very common. These seem to cause surprisingly few clinical problems. However, it should be noted that several of the actual symptoms that CVC-related thrombosis can cause may go unnoticed or misinterpreted as symptoms of the disease that caused the patient's to need of a CVC. It is important to know the true incidence of subclinical CVC-related thrombosis in order to evaluate the risk-benefit of central venous access compared to alternatives (peripheral venous access, midline, PICCLINE, porth-a-cath), and in the development of new less thrombogenic CVC materials.

ELIGIBILITY:
Substudy 1

Inclusion Criteria:

* Diseased patients with an indwelling central venous catheter and a clinical indication for autopsy
* Informed and signed consent from next of kind

Exclusion Criteria:

* None

Substudy 2 Inclusion Criteria

* Living patients with an indwelling central venous catheter who are referred to a CT scan without iv contrast
* Informed and signed consent from the patient

Exclusion Criteria

- GFR <15 mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Substudy 1: Diseased patients with an indwelling central venous catheter and a clinical indication for autopsy
  Substudy 2: Living patients with an indwelling central venous catheter who are referred to a CT scan without iv contrast
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of venous thrombosis related to a central venous catheter in diseased patients | At autopsy
  Venous thrombosis related to a central venous catheter detected at autopsy
The performance of the photon counting CT on diseased patients | After death. The CT scan and the autopsy will be performed within 1 week after death
  The performance of the photon counting CT will be evaluated by comparing the findings from the CT with the findings from the autopsy
The incidence of venous thrombosis related to a central venous catheter in living patients | At CT scan
  The incidence of venous thrombosis related to a central venous catheter in living patients detected with a photon counting CT
The performance of ultrasound compared to the photon counting CT | Ultrasound will be performed ±24 hours from the CT
  The performance of ultrasound compared to the photon counting CT in detecting enous thrombosis related to central venous catheters

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, Principal Investigator — Lund University
Locations (1):
- Intensive and Perioperative Care. Skåne University Hospital. Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, de-identified individual participant data from this clinical trial will be shared to facilitate scientific collaboration.
Supporting Information: Study Protocol, CSR
Time Frame: After the publication of the study up to 3 years after the publication of the study
Access Criteria: Researchers may submit requests through the specified channel, detailing the purpose and proposed analyses. Approved applicants will sign a data access agreement, ensuring responsible and transparent use of the data.

REFERENCES:
- [Background] Forauer AR, Theoharis C. Histologic changes in the human vein wall adjacent to indwelling central venous catheters. J Vasc Interv Radiol. 2003 Sep;14(9 Pt 1):1163-8. doi: 10.1097/01.rvi.0000086531.86489.4c. PMID 14514808
- [Background] Wichmann D, Heinemann A, Zahler S, Vogel H, Hopker W, Puschel K, Kluge S. Prospective study of device-related complications in intensive care unit detected by virtual autopsy. Br J Anaesth. 2018 Jun;120(6):1229-1236. doi: 10.1016/j.bja.2018.02.031. Epub 2018 Apr 4. PMID 29793590
- [Background] Rockholt MM, Naddi L, Badri AM, Englund E, Kander T. Macro- and microscopic changes in veins with short-term central venous catheters: an observational autopsy study. BMC Anesthesiol. 2024 Jan 2;24(1):5. doi: 10.1186/s12871-023-02380-x. PMID 38166620